CLINICAL TRIAL: NCT05533372
Title: Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of IA-14069 in Healthy Subjects, With an Extension to Explore Any Drug-Drug Interaction Potential With Methotrexate (Part 1), and in Patients With Rheumatoid Arthritis, With Preliminary Assessment of Efficacy in Patients (Part 2)
Brief Title: MAD Study of IA-14069
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ILAb Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: IA-14069_1b
Record Dates: First submitted 2022-09-05; First posted 2022-09-09 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- IA-14069 MAD (Experimental): Subjects will be administrated multiple oral doses of IA-14069 at three ascending dose levels or matching placebo for 10 days.
  Interventions: Drug: IA-14069; Drug: Placebo
- IA-14069 DDI (Experimental): Subjects will be administrated multiple oral doses of IA-14069 at three ascending dose levels or matching placebo for 10 days.
  On day 11, subjects will be adminiatrated oral dose of IA-14069 or matching placebo with methotrexate.
  On day 21, subjects will be administrated methotrexate alone.
  Interventions: Drug: IA-14069; Drug: Placebo; Drug: Methotrexate
- IA-14069 MAD RA patients (Experimental): Patients will be administrated multiple oral doses of IA-14069 at three ascending dose levels or matching placebo for 28 days.
  Patients will be on a stable dose of methotrexate throughout the study period.
  Interventions: Drug: IA-14069; Drug: Placebo; Drug: Methotrexate

INTERVENTIONS:
Drug: IA-14069 — IA-14069 for oral administration.
Drug: Placebo — Placebo for oral administration.
Drug: Methotrexate — Methotrexate for oral or SC administration.
  Arms: IA-14069 MAD RA patients
Drug: Methotrexate — Methotrexate for oral administration.
  Arms: IA-14069 DDI

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple ascending oral doses of IA-14069 in healthy subjects and in patients with RA on stable dosese of MTX, with preliminary assessment of efficacy in RA patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sex : Males or females; females may be of childbearing potential, of nonchildbearing potential, or postmenopausal.
2. Age : 18 to 55 years, inclusive, for healthy subjects in Part 1 and 18 to 70 years, inclusive, for RA patients in Part 2, at screening.
3. Body mass index (BMI) : 18 to 32 kg/m2, inclusive, for healthy subjects in Part 1 and 18 to 40 kg/m2, inclusive, for RA patients in Part 2, at screening.
4. Weight : ≥ 50 kg, inclusive, at screening.
5. Status : Healthy subjects for Part 1 and RA patients for Part 2.
6. At screening, females must not be pregnant or lactating.
7. At screening, females may be of nonchildbearing potential, either surgically sterilized, physiologically incapable of becoming pregnant, or postmenopausal.
8. Female subjects/patients of childbearing potential who have a fertile male sexual partner (ie, not surgically sterilized for at least 6 months prior to screening) must agree to use adequate contraception from at least 4 weeks prior to administration of the study drug until 90 days after the last dosing of study drug.
9. Male subjects/patients, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from admission to the clinical site until 90 days after the last dosing of study drug.
10. Non-use of all over-the-counter medication, vitamin preparations and other food supplements, or herbal medications (eg, St. John's wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) before administration of study drug until completion of the follow-up assessment, unless, judged by the Investigator in consultation with the Medical Monitor and the Sponsor that the medication will not interfere with the study drug.
11. Ability and willingness to abstain from alcohol from 72 hours (3 days) prior to each admission to the clinical site and until discharge.

    For North America only: Ability and willingness to abstain from caffeine, and methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, or energy drinks) from 72 hours (3 days) prior to each admission to the clinical site and until discharge.

    For EU only: Ability and willingness to abstain from caffeine, and methylxanthine-containing beverages or food (coffee, tea, cola, chocolate, or energy drinks) from 48 hours (2 days) prior to each admission to the clinical site and until discharge.
12. Good physical and mental health on the basis of medical history (except for RA medical history in Part 2 of the study), physical examinations, clinical laboratory tests, 12-lead ECG, and vital signs, as judged by the Investigator.
13. Resting supine blood pressure showing no clinically relevant deviations as judged by the Investigator. If initial results do not meet these criteria, blood pressure and/or pulse may be repeated if in the judgment of the Investigator there is a reason to believe the initial result is inaccurate (eg, white coat hypertension).
14. Computerized 12-lead ECG recording without signs of clinically relevant pathology or showing no clinically relevant deviations as judged by the Investigator. The ECG may be repeated if in the judgment of the Investigator there is a reason to believe the initial result is inaccurate.
15. All values for clinical laboratory tests of blood and urine within the normal range or showing no clinically relevant deviations as judged by the Investigator. Clinical laboratory tests may be repeated at the discretion of the Investigator.
16. Willing and able to sign the ICF.

    Main inclusion criteria; Part 2 in RA patients only:
17. Treatment with oral or SC MTX 5 to 25 mg QW as a DMARD for at least 12 weeks prior to screening, and with a stable oral or SC dose for at least 4 weeks before screening, and that is expected to remain stable throughout the study period.
18. Having active RA, defined as:

    * at least 6 swollen and 6 tender joints (based on 66/68 joint count), and
    * CRP ≥ ULN or ESR ≥ ULN

Exclusion Criteria:

1. Previous participation in the SAD study (Study IA-14069_1a).
2. Employee of ICON or the Sponsor.
3. Use of any investigational drug or device within 30 days (or 5 half-lives if known, whichever is longer) prior to admission.
4. Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the subjects or patients.
5. Females who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the last dosing of study drug.
6. Males with female partners who are pregnant, lactating, or planning to attempt to become pregnant during this study or within 90 days after the last dosing of study drug.
7. History of relevant drug sensitivity, and/or food allergies, as determined by the Investigator (such as anaphylaxis, hepatotoxicity, or treatment with steroids or epinephrine). Confirmatory circumstances would include treatment with epinephrine or in Emergency Department.
8. Allergy or hypersensitivity to active ingredient or excipients.
9. Using tobacco or nicotine products within 60 days prior to study drug administration (for subjects in Part 1).
10. History within the previous 12 months of alcohol consumption exceeding 2 standard drinks per day on average (1 standard drink=12 oz beer, 5 oz wine, and 1.5 oz spirits).
11. Positive drug and alcohol screen (opiates, methadone, cocaine, amphetamines [including ecstasy], phencyclidine, cannabinoids, barbiturates, benzodiazepines, tricyclic antidepressants, cotinine [only exclusionary in Part 1], and alcohol) at screening or admission to the clinical site.
12. Positive screen for hepatitis B surface antigen (HbsAg), hepatitis C virus (HCV) antibodies, or HIV-1 and -2 antibodies.
13. Donation or loss of more than 450 mL of blood within 60 days prior to study drug administration, or planned donation before 30 days has elapsed after the last dosing of study drug.
14. Plasma or platelet donation within 7 days prior to study drug administration through follow-up assessment.
15. Significant and/or acute illness within 5 days prior to drug administration that may impact safety assessments, in the opinion of the Investigator.
16. Unsuitable veins for blood sampling.
17. Chronic use of prescription or nonprescription drugs (including vitamins and dietary or herbal supplements) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives if known (whichever is longer) prior to the first dosing (except oral or SC MTX, oral glucocorticoid [prednisone ≤ 10 mg/day or equivalent; this exception is allowed if stable for at least 3 months prior to screening and expected to remain stable throughout the study period], folic acid and/or folinic acid in Part 2), but considered on a case-by-case basis by the Investigator in consultation with the Medical Monitor and the Sponsor.
18. Patients receiving a biologic DMARD, or having received a biologic DMARD within 6 weeks or 5 half-lives if known (whichever is longer) prior to screening (Part 2 only).
19. Patients receiving a targeted synthetic DMARD (including apremilast, baricitinib, filgotinib, or tofacitinib), or having received a targeted synthetic DMARD within 6 weeks or 5 half-lives (whichever is longer) prior to screening (Part 2 only).
20. Patients receiving a conventional synthetic DMARD (except MTX), or having received a conventional synthetic DMARD within 6 weeks or 5 half-lives (whichever is longer) prior to screening (Part 2 only).
21. Strenuous activity, sunbathing, and contact sports within 48 hours (2 days) prior to admission to the clinical site through follow-up assessment.
22. Consumption of any nutrients known to modulate CYP enzymes activity (eg, grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) within 14 days prior to administration of study drug and during the study.
23. Unable to comply with the safety monitoring requirements of this clinical study or is considered by the Investigator to be an unsuitable candidate for the study.
24. Received a SARS-CoV-2 or any other vaccine within 7 days prior to dosing of study drug.

    Main exclusion criteria; Part 1 in healthy subjects only:
25. Clinically significant hepatic impairment demonstrated by ALT, AST, total bilirubin, gamma-glutamyl transferase (GGT), and prothrombin time as judged by the Investigator at screening and on Day -1.
26. Clinically significant renal impairment evidenced by estimated glomerular filtration rate (eGFR) calculated with the Chronic Kidney Disease EpidemiologyCollaboration (CKD-EPI) 2021, and protein in urine as judged by the Investigator at screening and on Day -1.

    Main exclusion criteria; Part 2 in RA patients only:
27. Patients with any single parameter of ALT, AST, GGT, or alkaline phosphatase (ALP) exceeding 2.5×ULN or total bilirubin exceeding 1.5×ULN OR any elevation above ULN of more than one parameter of ALT, AST, GGT, ALP, or serum bilirubin at screening and on Day -3.
28. Patients with eGFR value calculated with the CKD-EPI 2021 <60 mL/min/1.73m2 at screening and on Day -3.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Incidnece and severity of adverse events | up to Day 35
  Incidence and severity of adverse events (AEs) and serious AEs, including clinical laboratory values, vital signs, 12-lead electrocardiograms, and physical examination; changes from baseline.

SECONDARY OUTCOMES:
Cmax | up to Day 28
  Maximum ovserved plasma concentration of IA-14069 and/or methotrexate
Tmax | up to Day 28
  Time to attain maximum observed plasma concentration of IA-14069 and/or methotrexate
AUC | up to Day 28
  Area under the plasma concentration time curve of IA-14069 and/or methotrexate
t1/2el | up to Day 28
  Terminal elimination half-life of IA-14069 and/or methotrexate
CL/F | up to Day 28
  Apparent clearance (CL/F) of IA-14069
VD/F | up to Day 28
  Apparent volume of distribution (Vd/F) of IA-14069

OTHER OUTCOMES:
Change from baseline in concentration of Tumor necrosis factor in blood | up to Day 28
Change from baseline in disease activity scores | up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- ICON plc., Lenexa, Kansas, United States